CLINICAL TRIAL: NCT06225011
Title: Repurposing Drugs as Immunotherapeutic Agents: Changes in Colorectal Tumor Immune Cells After Targeting Serotonin
Brief Title: Fluoxetine for the Modification of Colorectal Tumor Immune Cells Before Surgery in Patients With Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-001744; NCI-2023-09939 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-01-04; First posted 2024-01-25 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Adenocarcinoma
MeSH Terms: interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (fluoxetine) (Experimental): Patients receive fluoxetine PO once QD for 10 days prior to surgery.
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine — Receive PO

SUMMARY:
This phase I trial tests whether fluoxetine (prozac) works to modify the tumor immune cells before surgery in patients with colorectal cancer. Fluoxetine is a commonly used selective serotonin reuptake inhibitor (SSRI) prescribed for major depressive disorder and generalized anxiety. Giving fluoxetine may modify the immune cell composition in the tumor and its microenvironment and may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread in patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate alterations in tumor immune cell composition and activity under SSRI treatment.

OUTLINE:

Patients receive fluoxetine orally (PO) once daily (QD) for 10 days prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age at visit 1
* Previously untreated cytologically or histologically confirmed colorectal adenocarcinoma that will not need neoadjuvant therapy
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study
* World Health Organization (WHO) Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1.5x10^9/L
* Platelets ≥ 100x10^9/L
* Hemoglobin ≥ 9 g/dL
* Serum creatinine (sCr) ≤ 1.5 x upper limit of normal (ULN)
* Creatinine clearance (Ccr) ≥ 40 mL/min (as calculated by Modified Cockcroft-Gault formula)
* Serum total bilirubin ≤ 1.5 x ULN
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 x ULN
* Baseline corrected QT (QTc) within normal limits per the Bazett formula. Any electrocardiogram (EKG) done prior to consent is acceptable for baseline QTc monitoring.

  * Normal QTc ranges from 350-450 ms for adult men and from 360-460 ms for adult women

Exclusion Criteria:

* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the participant or the quality of the data
* A diagnosis of metastatic colorectal adenocarcinoma
* Individuals who have received neoadjuvant chemotherapy prior to the planned colon cancer resection
* Individuals with absolute or relative contraindications to fluoxetine

  * Baseline prolonged QTc
  * Concurrently taking tamoxifen, pimozide, or thioridazine
* Individuals using other SSRIs, serotonin and norepinephrine reuptake inhibitors (SNRIs), monoamine oxidase inhibitors (MAOIs), lithium or other antidepressants at time of initial biopsy
* Currently active second primary malignancy or history of malignancy less than 5 years prior to the time of study eligibility (Patients with history of skin cancers excluding melanoma will be eligible for participation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Immune cell composition and microenvironment | within a year of surgery
  Will be assessed by changes in the immune cell composition in the tumor and its microenvironment before and after exposure to selective serotonin reuptake inhibitors therapy. Fixed tumor samples will be analyzed by immunohistochemistry for immune cell tumor infiltration and relevant lineage/activation/exhaustion markers. Will use descriptive statistics and graphical displays to compare the changes in tumor immune markers between the pre- and post-treatment tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine Mitchell, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States